CLINICAL TRIAL: NCT05801315
Title: Treatment of Peri-implant Mucositis: Adjunctive Benefit of Glycine Powder Air Polishing Device to Professional Mechanical Biofilm Removal. A Randomized Parallel Arm Clinical Study
Brief Title: Non-surgical Treatment of Peri-implant Mucositis: FMUD vs FMUD and Air-Flow Master Piezon®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Nicola Discepoli, Professor, University of Siena
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MU001
Record Dates: First submitted 2020-03-04; First posted 2023-04-06 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Peri-implant Mucositis
Keywords: Peri-implant Mucosits; air polishing device; non-surgical treatment

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Full mouth ultrasonic debridement plus glycine powder air polishing (Experimental): Plaque and calculus are firstly removed through full mouth ultrasonic debridement (FMUD) in all sites (both dental and implant). After this procedure an air polishing device (Air-flow Master Piezon®) is used as additional therapy to further debride peri-implant trans-mucosal tract.
  Interventions: Device: Glycine powder air polishing; Device: Full mouth ultrasonic debridement
- Full mouth ultrasonic debridement (Active Comparator): Plaque and calculus are removed through full mouth ultrasonic debridement (FMUD) in all sites (both dental and implant).
  Interventions: Device: Full mouth ultrasonic debridement

INTERVENTIONS:
Device: Glycine powder air polishing — Peri-implant mucositis sites treated with a glycine powder air polishing device (Air-Flow Master Piezon®).
  Arms: Full mouth ultrasonic debridement plus glycine powder air polishing
Device: Full mouth ultrasonic debridement — Peri-implant mucositis sites are treated with thin ultrasonic tips.

SUMMARY:
The aim of the present study is to evaluate the adjunctive effect of glycine-powder air-polishing (GPAP) to full-mouth ultrasonic debridement (Fm-UD) in the treatment of peri-implant mucositis, and to determine the predictive role of implant and patient-level variables for disease resolution. Both treatments are described in the literature, but few studies are available on their comparison.

DETAILED DESCRIPTION:
52 patients (132 implants) with peri-implant mucositis were included in this randomized parallel arm clinical study. Following baseline variables assessment, participants received Fm-UD. Implants allocated to the test group (n=64) were additionally treated with GPAP. Clinical outcomes were evaluated at 3 and 12 months following intervention. Complete and partial disease resolution were defined as absence of BoP (DR1) or <2 BoP+ sites (DR2), respectively.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 70 years old;
* presence of one implant loaded at least one year before;
* bleeding on probing and/or suppuration of the peri-implant mucosa;
* pain and/or tenderness of the peri-implant mucosa;
* good general health conditions.

Exclusion Criteria:

* radiographic bone loss ≥ 2mm;
* intake of anticoagulants, antiplatelet, antibiotic or cortisone drugs;
* inability to perform oral hygiene maneuvers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Bleeding on probing | 12 months
  After probing dental and implant sites a dichotomic value (0/1) is assigned for each site. 0: not bleeding site; 1: bleeding site.

SECONDARY OUTCOMES:
Probing pocket depth change | 12 months
  Change in probing pocket depth measured in millimeter through a periodontal probe.

CONTACTS AND LOCATIONS:
Locations (1):
- AOUS, Siena, Italy

REFERENCES:
- [Derived] Nicola D, Isabella R, Carolina C, Baldini N, Raffaele M. Treatment of peri-implant mucositis: Adjunctive effect of glycine powder air polishing to professional mechanical biofilm removal. 12 months randomized clinical study. Clin Implant Dent Relat Res. 2024 Apr;26(2):415-426. doi: 10.1111/cid.13304. Epub 2024 Feb 5. PMID 38317375